CLINICAL TRIAL: NCT02969044
Title: A Phase 2a, Randomized, Double-blind, Parallel Group, Placebo-controlled, Multi-center Study To Assess The Efficacy And Safety Profile Of Pf-06651600 In Subjects With Moderate To Severe Active Rheumatoid Arthritis With An Inadequate Response To Methotrexate
Brief Title: Study To Assess The Efficacy And Safety Of Pf-06651600 In Subjects With Rheumatoid Arthritis With An Inadequate Response To Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981006; 2016-002862-30 (EudraCT Number)
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — PF-06651600

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-06651600 (Experimental): Study Drug
  Interventions: Drug: PF-06651600
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: PF-06651600 — 200mg pill every day (QD) for 8 weeks
  Arms: PF-06651600

SUMMARY:
This is an 8 week study to assess the efficacy and safety profile of PF-06651600 in seropositive subjects with rheumatoid arthritis with an inadequate response to methotrexate (up to approximately 50% of subjects may also have had an inadequate response to 1 anti-TNF biologic).

ELIGIBILITY:
Inclusion Criteria

* Subjects between the ages of 18 and 75 years, inclusive
* Must have moderate-to-severe, active Rheumatoid Arthritis
* Must have had an inadequate response to Methotrexate
* Subjects may have received one approved TNF inhibiting biologic agent that was inadequately effective and/or not tolerated

Exclusion Criteria

* Subjects with any acute or chronic infections or infection history
* Have acute or active chronic dermatological disorders prior to study start
* Any major illness/condition(s) or evidence of an unstable clinical condition that in the judgment of the investigator would make the subject inappropriate for entry into this study
* Known immunodeficiency disorder or a first degree relative with hereditary immunodeficiency
* Any live (attenuated) vaccines or current routine household contact with anyone who has received live (attenuated) vaccine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (4):
  - California Medical Research Associates Inc., Northridge, California
  - Clayton Medical Associates, PC, St Louis, Missouri
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
- Bulgaria (5):
  - MHAT "Trimontsium" Department of Internal Diseases, Plovdiv
  - UMHAT Kaspela, Clinic of Rheumatology, Plovdiv
  - Medical Centre "Pirogov", Sofia
  - Medical Center Equita, Varna
  - Medical Center "Sveti Ivan Rilski", Vidin
- MEDICAL PLUS, s.r.o., Uherské Hradiště, Czechia
- Georgia (4):
  - LTD "Unimed Ajara" Batumi Referral Hospital, Batumi
  - LTD Israeli-Georgian Medical Research Clinic ,,Helsicore", Tbilisi
  - Ltd Institute of Clinical Cardiology, Tbilisi
  - LTD Unimedi Kakheti, Tbilisi
- Germany (2):
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Rheumatologische Schwerpunktpraxis, Berlin
- Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Klinikai Kutatasi Osztaly, Nyíregyháza, Hungary
- Poland (5):
  - NZOZ Centrum Medyczne Sw. Lukasza w Kartuzach, Kartuzy
  - Care Clinic Sp. z o.o., Katowice
  - Silmedic Sp. z o.o. Oddzial w Katowicach, Katowice
  - Oswiecimskie Centrum Badan Klinicznych Medicome Sp. z o.o., Oświęcim
  - Centrum Medyczne Oporow, Wroclaw
- Serbia (4):
  - Clinic of Dermatovenerology "Prof. Zecevic", Belgrade
  - Institute of Rheumatology, Belgrade
  - Polyclinic Medikom, Belgrade
  - Institute of Treatment and Rehabilitation "Niska Banja", Niška Banja
- Slovakia (4):
  - AAGS s.r.o., Reumatologicka ambulancia, Dunajská Streda
  - MUDr. Zuzana Cizmarikova s.r.o. , Reumatologicka ambulancia, Poprad
  - Nestatna reumatologicka ambulancia, Považská Bystrica
  - Reumatologicka ambulancia, MUDr. Pavol Polak s.r.o., Žilina

REFERENCES:
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- [Derived] Purohit V, Huh Y, Wojciechowski J, Plotka A, Salts S, Antinew J, Dimitrova A, Nicholas T. Leveraging Prior Healthy Participant Pharmacokinetic Data to Evaluate the Impact of Renal and Hepatic Impairment on Ritlecitinib Pharmacokinetics. AAPS J. 2023 Mar 28;25(3):32. doi: 10.1208/s12248-023-00792-8. PMID 36977960
- [Derived] Robinson MF, Damjanov N, Stamenkovic B, Radunovic G, Kivitz A, Cox L, Manukyan Z, Banfield C, Saunders M, Chandra D, Vincent MS, Mancuso J, Peeva E, Beebe JS. Efficacy and Safety of PF-06651600 (Ritlecitinib), a Novel JAK3/TEC Inhibitor, in Patients With Moderate-to-Severe Rheumatoid Arthritis and an Inadequate Response to Methotrexate. Arthritis Rheumatol. 2020 Oct;72(10):1621-1631. doi: 10.1002/art.41316. Epub 2020 Sep 7. PMID 32419304
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981006&StudyName=A+Phase+2a%2C+Randomized%2C+Double-blind%2C+Parallel+Group%2C+Placebo-controlled%2C+Multi-center+Study+To+Assess+The+Efficacy+And+Safety+Profile+Of+Pf-06651600+In+Subjects+With+Moderate+To+Severe+Active+Rheumatoid+Arthritis+With+An+Inadequate+Response+To+Methotrexate
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981006&StudyName=A+Phase+2a%2C+Randomized%2C+Double-blind%2C+Parallel+Group%2C+Placebo+Controlled%2C+Multi-center+Study+To+Assess+The+Efficacy+And+Safety+Profile+Of+Pf-06651600+In+Subjects+With+Moderate+To+Severe+Active+Rheumatoid+Arthritis+With+An+Inadequate+Response+To+Methotrexate

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06651600: Participants received 200 milligram (mg) of PF-06651600 tablet once daily for a period of 8 weeks. Participants were followed up to 4 weeks after last dose of investigational drug.
- Placebo: Participants received placebo matched to 200 mg of PF-06651600 tablet once daily for a period of 8 weeks. Participants were followed up to 4 weeks after last dose of investigational drug.
Period: Overall Study
Arm/Group | PF-06651600 | Placebo
Started | 42 | 28
Completed | 37 | 22
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all participants who were randomized to the study and received at least one dose of the randomized investigational drug (PF-06651600 or placebo).
Groups:
- PF-06651600: Participants received 200 mg of PF-06651600 tablet once daily for a period of 8 weeks. Participants were followed up to 4 weeks after last dose of investigational drug.
- Total: Total of all reporting groups
Arm/Group | PF-06651600 | Placebo | Total
Number analyzed (Participants) | 42 | 28 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (11.72) | 54.2 (11.78) | 54.9 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 24 | 57
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 41 | 26 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 41 | 28 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Simple Disease Activity Index (SDAI) Score at Week 8
Description: The SDAI is the numerical sum of five outcome parameters: tender joint count (TJC) and swollen joint count (SJC) based on a 28-joint assessment, patient global assessment (PtGA) and physician global assessment (PGA) assessed on a visual analogue scale (VAS) scale ranging from 0 to 10 centimeter (cm), where higher scores=greater affection due to disease activity, and C-reactive protein (CRP) measured in terms of milligram per deciliter (mg/dL). SDAI total score= 0 to 86. SDAI greater than or equal to (<=) 3.3 indicates disease remission, greater than (>) 3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Time Frame: Baseline, Week 8
Population: ITT analysis set included all participants who were randomized to the study and received at least one dose of the randomized investigational drug (PF-06651600 or placebo). Here, n signifies number of participants evaluable at specified time points only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
units on a scale
  Baseline | 45.15 (13.164) | 44.85 (13.976)
  Change at Week 8: number analyzed (Participants) | 39 | 24
  Change at Week 8 | -26.11 (14.834) | -17.38 (18.176)
Statistical Analysis 1: Comparison: PF-06651600 vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -9.25, 95% CI 2-sided [-14.75 to -3.79]

2. Secondary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Criteria: sitting pulse rate less than (<) 40 beats per minute (bpm) or >120 bpm; sitting systolic blood pressure (SBP) >=30 millimeters of mercury (mmHg) change from baseline in same posture or <90 mmHg; diastolic blood pressure (DBP) >=20 mmHg change from baseline in same posture or <50 mmHg. Only those categories in which at least one participant had abnormality, were reported in this outcome measure.
Time Frame: Baseline up to Week 12
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
Participants
  Sitting DBP >=20 mmHg increase from baseline | 3 | 0
  Sitting DBP >=20 mmHg decrease from baseline | 0 | 1

3. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Hemoglobin(Hb);hematocrit;RBC count:<0.8*lower limit of normal (LLN),mean corpuscular volume;mean corpuscular Hb concentration:<0.9*LLN or>1.1*upper limit of normal (ULN), platelet:<0.5*LLN or >1.75*ULN,reticulocytes <0.5*LLN or >1.5*ULN,leukocytes <0.6*LLN or >1.5*ULN,lymphocyte;neutrophil: <0.8*LLN or >1.2*ULN,basophil;eosinophil; monocyte:>1.2*ULN,partial thromboplastin time,prothrombin time>1.1*ULN,bilirubin>1.5*ULN, aspartate aminotransferase; alanine aminotransferase;alkaline phosphatase:>3.0*ULN,protein;albumin;LDL, HDL cholesterol:<0.8*LLN or >1.2*ULN;urea nitrogen;creatinine: >1.3*ULN, urate >1.2*ULN, sodium<0.95*LLN or >1.05*ULN, potassium; chloride;calcium; bicarbonate:<0.9*LLN or >1.1*ULN,glucose <0.6*LLN or >1.5*ULN, creatine kinase: >2.0*ULN;urine pH <4.5 or >8,urine glucose or ketones>=1,urine protein;urineHb>=1,urobilinogen;bilirubin;nitrite;leukocyte esterase >=1,urine erythrocytes, leukocytes>=20,hyaline cast>1,bacteria>20.
Time Frame: Baseline up to Week 12
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
Participants | 42 | 28

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 12 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Week 12
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
Participants
  AEs | 20 | 5
  SAEs | 0 | 0

5. Secondary Outcome: Change From Baseline in Simple Disease Activity Index (SDAI) Score at Week 1, 2, 4 and 6
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on a VAS scale ranging from 0 to 10 cm, where higher scores=greater affection due to disease activity, and CRP measured in terms of mg/dL. SDAI total score= 0 to 86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Time Frame: Baseline, Week 1, 2, 4 and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
units on a scale
  Change at Week 1: number analyzed (Participants) | 40 | 28
  Change at Week 1 | -4.59 (9.409) | -4.52 (7.025)
  Change at Week 2: number analyzed (Participants) | 42 | 27
  Change at Week 2 | -12.82 (10.969) | -8.05 (9.402)
  Change at Week 4: number analyzed (Participants) | 41 | 26
  Change at Week 4 | -17.79 (12.804) | -12.55 (13.462)
  Change at Week 6: number analyzed (Participants) | 40 | 26
  Change at Week 6 | -22.79 (14.007) | -15.62 (14.231)

6. Secondary Outcome: Remission Rate Based on Simple Disease Activity Index Score
Description: Remission rate was defined as percentage of participants with disease remission. The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on a VAS scale ranging from 0 to 10 cm, where higher scores=greater affection due to disease activity, and CRP measured in terms of mg/dL. SDAI total score= 0 to 86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Time Frame: Week 4, 6 and 8
Population: ITT analysis set included all participants who were randomized to the study and received at least one dose of the randomized investigational drug (PF-06651600 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
percentage of participants
  Week 4 | 4.8 | 0.0
  Week 6 | 4.8 | 0.0
  Week 8 | 7.1 | 0.0

7. Secondary Outcome: Remission Rate Based on Disease Activity Score (DAS28-3 [ESR])
Description: Remission rate was defined as the percentage of participants with disease remission. DAS28 is measure of disease activity in participants with rheumatoid arthritis. DAS28-3 (ESR) was calculated from SJC and TJC using 28 joints count, and erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]). Total score range: 0-9.4, higher score=more disease activity. DAS28-3 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (ESR) <2.6 = remission.
Time Frame: Week 4, 6 and 8
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
percentage of participants
  Week 4 | 4.8 | 0.0
  Week 6 | 2.4 | 0.0
  Week 8 | 7.1 | 0.0

8. Secondary Outcome: Remission Rate Based on Disease Activity Score (DAS28-4[ESR])
Description: Remission rate was defined as the percentage of participants with disease remission. DAS28 is measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from the number of SJC and TJC using the 28 joints count, the ESR (mm/hour) and participant's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). Total score range: 0-9.4, higher score=more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) <2.6 = remission.
Time Frame: Week 4, 6 and 8
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
percentage of participants
  Week 4 | 4.8 | 0.0
  Week 6 | 4.8 | 0.0
  Week 8 | 7.1 | 0.0

9. Secondary Outcome: Remission Rate Based on Disease Activity Score (DAS28-3 [CRP])
Description: Remission rate was defined as the percentage of participants with disease remission. DAS28 is measure of disease activity in participants with rheumatoid arthritis. DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Week 4, 6 and 8
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
percentage of participants
  Week 4 | 9.5 | 0.0
  Week 6 | 7.1 | 3.6
  Week 8 | 9.5 | 0.0

10. Secondary Outcome: Remission Rate Based on Disease Activity Score (DAS28-4 [CRP])
Description: Remission rate was defined as the percentage of participants with disease remission. DAS28 is measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP): calculated from SJC, TJC, CRP (mg/L) and PGA (participant rated disease activity on VAS from 0 to 100 mm; high score=worse health). Total score range of DAS28-4 (CRP): 0 to 9.4(0=no activity; 9.4=extreme disease activity), higher score=more disease activity. DAS28-4(CRP) <2.6=remission, <3.2=low disease activity, >=3.2-5.1=moderate disease activity and >5.1=high disease activity.
Time Frame: Week 4, 6 and 8
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
percentage of participants
  Week 4 | 9.5 | 0.0
  Week 6 | 9.5 | 3.6
  Week 8 | 9.5 | 0.0

11. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (3 Variables) (DAS28-3 [ESR]) at Week 1, 2, 4, 6 and 8
Description: DAS28 is measure of disease activity in participants with rheumatoid arthritis. DAS28-3 (ESR) was calculated from SJC and TJC using 28 joints count, and ESR (mm/hr). Total score range: 0-9.4, higher score=more disease activity. DAS28-3 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (ESR) <2.6 = remission.
Time Frame: Baseline, Week 1, 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
units on a scale
  Baseline | 6.49 (0.762) | 6.37 (0.815)
  Change at Week 1: number analyzed (Participants) | 40 | 28
  Change at Week 1 | -0.19 (0.604) | -0.26 (0.434)
  Change at Week 2: number analyzed (Participants) | 42 | 27
  Change at Week 2 | -0.67 (0.602) | -0.46 (0.531)
  Change at Week 4: number analyzed (Participants) | 41 | 26
  Change at Week 4 | -1.16 (1.125) | -0.78 (0.905)
  Change at Week 6: number analyzed (Participants) | 40 | 25
  Change at Week 6 | -1.54 (1.123) | -1.07 (0.989)
  Change at Week 8: number analyzed (Participants) | 39 | 24
  Change at Week 8 | -1.85 (1.161) | -1.07 (1.214)

12. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Week 1, 2, 4, 6 and 8
Description: DAS28 is measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hr) and PtGA of disease activity (participant rated arthritis activity assessment). Total score range: 0-9.4, higher score=more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) <2.6 = remission.
Time Frame: Baseline, Week 1, 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
units on a scale
  Baseline | 6.82 (0.815) | 6.72 (0.880)
  Change at Week 1: number analyzed (Participants) | 40 | 28
  Change at Week 1 | -0.27 (0.553) | -0.27 (0.477)
  Change at Week 2: number analyzed (Participants) | 42 | 27
  Change at Week 2 | -0.83 (0.695) | -0.47 (0.551)
  Change at Week 4: number analyzed (Participants) | 41 | 26
  Change at Week 4 | -1.36 (1.173) | -0.89 (0.951)
  Change at Week 6: number analyzed (Participants) | 40 | 25
  Change at Week 6 | -1.81 (1.179) | -1.18 (1.050)
  Change at Week 8: number analyzed (Participants) | 39 | 24
  Change at Week 8 | -2.14 (1.269) | -1.22 (1.448)

13. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Week 1, 2, 4, 6 and 8
Description: DAS28 is measure of disease activity in participants. DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Baseline, Week 1, 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
units on a scale
  Baseline | 5.76 (0.824) | 5.61 (0.894)
  Change at Week 1: number analyzed (Participants) | 40 | 28
  Change at Week 1 | -0.35 (0.741) | -0.20 (0.456)
  Change at Week 2: number analyzed (Participants) | 42 | 27
  Change at Week 2 | -0.86 (0.782) | -0.47 (0.585)
  Change at Week 4: number analyzed (Participants) | 41 | 26
  Change at Week 4 | -1.33 (1.219) | -0.72 (1.005)
  Change at Week 6: number analyzed (Participants) | 40 | 26
  Change at Week 6 | -1.53 (1.286) | -1.01 (0.993)
  Change at Week 8: number analyzed (Participants) | 39 | 24
  Change at Week 8 | -1.79 (1.265) | -1.03 (1.146)

14. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (4 Variables) (DAS28-4 [CRP]) at Week 1, 2, 4, 6 and 8
Description: DAS28 is measure of disease activity in participants. DAS28-4 (CRP): calculated from SJC, TJC, CRP(mg/L) and PGA (participant rated disease activity on VAS from 0 to 100 mm; high score=worse health). Total score range of DAS28-4 (CRP): 0 to 9.4(0=no activity; 9.4=extreme disease activity), higher score=more disease activity. DAS28-4(CRP) <2.6=remission, <3.2=low disease activity, >=3.2-5.1=moderate disease activity and >5.1=high disease activity.
Time Frame: Baseline, Week 1, 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
units on a scale
  Baseline | 6.11 (0.850) | 5.98 (0.926)
  Change at Week 1: number analyzed (Participants) | 40 | 28
  Change at Week 1 | -0.41 (0.685) | -0.21 (0.473)
  Change at Week 2: number analyzed (Participants) | 42 | 27
  Change at Week 2 | -0.99 (0.823) | -0.47 (0.574)
  Change at Week 4: number analyzed (Participants) | 41 | 26
  Change at Week 4 | -1.49 (1.222) | -0.82 (1.013)
  Change at Week 6: number analyzed (Participants) | 40 | 26
  Change at Week 6 | -1.78 (1.304) | -1.09 (1.057)
  Change at Week 8: number analyzed (Participants) | 39 | 24
  Change at Week 8 | -2.06 (1.321) | -1.16 (1.367)

15. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP) Concentration at Week 1, 2, 4, 6 and 8
Time Frame: Baseline, Week 1, 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
milligram per deciliter
  Baseline | 2.00 (1.816) | 1.68 (2.853)
  Change at Week 1: number analyzed (Participants) | 40 | 28
  Change at Week 1 | -0.20 (2.672) | 0.60 (2.263)
  Change at Week 2: number analyzed (Participants) | 42 | 27
  Change at Week 2 | -0.62 (2.090) | -0.04 (0.966)
  Change at Week 4: number analyzed (Participants) | 41 | 26
  Change at Week 4 | -0.93 (1.591) | 0.00 (1.335)
  Change at Week 6: number analyzed (Participants) | 40 | 26
  Change at Week 6 | -0.42 (2.376) | -0.23 (1.327)
  Change at Week 8: number analyzed (Participants) | 39 | 24
  Change at Week 8 | -0.89 (2.142) | -0.04 (2.220)

16. Secondary Outcome: Change From Baseline in the Tender Joint Count and Swollen Joint Count at Week 1, 2, 4, 6 and 8
Description: Tender joint count was an assessment of 68 joints (upper body, upper extremity, and lower extremity). Each joint's response to pressure/motion was assessed as: Present or Absent. Swollen joint count was an assessment of 66 joints (upper body, upper extremity, and lower extremity). Each joint was assessed for swelling as: Present or Absent.
Time Frame: Baseline, Week 1, 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
joint count
  Baseline: Tender joint count | 16.74 (6.765) | 16.75 (6.681)
  Baseline: Swollen joint count | 12.95 (5.396) | 12.11 (6.160)
  Change at Week 1: Tender joint count: number analyzed (Participants) | 41 | 28
  Change at Week 1: Tender joint count | -1.54 (4.915) | -1.96 (2.701)
  Change at Week 1: Swollen joint count: number analyzed (Participants) | 41 | 28
  Change at Week 1: Swollen joint count | -1.49 (4.439) | -2.46 (3.501)
  Change at Week 2: Tender joint count: number analyzed (Participants) | 42 | 27
  Change at Week 2: Tender joint count | -4.40 (5.522) | -2.56 (5.213)
  Change at Week 2: Swollen joint count: number analyzed (Participants) | 42 | 27
  Change at Week 2: Swollen joint count | -4.71 (4.430) | -4.11 (4.619)
  Change at Week 4: Tender joint count: number analyzed (Participants) | 41 | 26
  Change at Week 4: Tender joint count | -6.76 (6.818) | -4.96 (7.750)
  Change at Week 4: Swollen joint count: number analyzed (Participants) | 41 | 26
  Change at Week 4: Swollen joint count | -5.95 (4.950) | -4.85 (4.961)
  Change at Week 6: Tender joint count: number analyzed (Participants) | 40 | 26
  Change at Week 6: Tender joint count | -8.75 (7.132) | -6.42 (6.652)
  Change at Week 6: Swollen joint count: number analyzed (Participants) | 40 | 26
  Change at Week 6: Swollen joint count | -7.80 (5.743) | -5.85 (5.540)
  Change at Week 8: Tender joint count: number analyzed (Participants) | 39 | 24
  Change at Week 8: Tender joint count | -10.21 (7.259) | -6.83 (7.755)
  Change at Week 8: Swollen joint count: number analyzed (Participants) | 39 | 24
  Change at Week 8: Swollen joint count | -8.59 (6.176) | -6.54 (6.324)

17. Secondary Outcome: Change From Baseline in Participant's Assessment of Arthritis Pain (PAAP), Participant's Global Assessment of Arthritis (PGA) and Physician's Global Assessment of Arthritis (PGAA) at Week 1, 2, 4, 6 and 8
Description: PAAP: Participants assessed the severity of their arthritis pain by using a 100 mm VAS ranging from 0 (no pain) to 100 (most severe pain), which corresponded to the magnitude of their pain, where higher scores indicated more pain. PGA: Participants were asked the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" and their response was recorded on a 100 mm VAS ranging from 0 (very well) to 100 (very poor), where higher scores indicated worse health condition. PGAA: Participants were assessed how their overall arthritis appears at the time of the visit. The evaluation was based on the participant's disease signs, functional capacity and physical examination, and was independent of the PAAP and PGA assessments. The physician's response was recorded using a 100 mm VAS ranging from 0 (very well) to 100 (very poor), where higher scores indicated more disease activity.
Time Frame: Baseline, Week 1, 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
units on a scale
  Baseline: PAAP | 66.64 (16.771) | 71.75 (16.183)
  Baseline: PGA | 68.43 (15.639) | 69.00 (16.115)
  Baseline: PGAA | 66.17 (14.228) | 74.07 (12.844)
  Change at Week 1: PAAP: number analyzed (Participants) | 41 | 28
  Change at Week 1: PAAP | -4.95 (11.388) | -2.86 (14.847)
  Change at Week 1: PGA: number analyzed (Participants) | 41 | 28
  Change at Week 1: PGA | -6.76 (11.128) | -1.93 (9.149)
  Change at Week 1: PGAA: number analyzed (Participants) | 41 | 28
  Change at Week 1: PGAA | -6.83 (8.947) | -4.96 (8.126)
  Change at Week 2: PAAP: number analyzed (Participants) | 42 | 27
  Change at Week 2: PAAP | -11.90 (18.061) | -6.04 (12.669)
  Change at Week 2: PGA: number analyzed (Participants) | 42 | 27
  Change at Week 2: PGA | -14.74 (15.963) | -2.81 (9.931)
  Change at Week 2: PGAA: number analyzed (Participants) | 42 | 27
  Change at Week 2: PGAA | -16.07 (16.499) | -10.63 (12.500)
  Change at Week 4: PAAP: number analyzed (Participants) | 41 | 26
  Change at Week 4: PAAP | -19.88 (16.695) | -10.23 (25.513)
  Change at Week 4: PGA: number analyzed (Participants) | 41 | 26
  Change at Week 4: PGA | -20.05 (13.746) | -12.12 (19.574)
  Change at Week 4: PGAA: number analyzed (Participants) | 41 | 26
  Change at Week 4: PGAA | -21.49 (16.715) | -17.96 (18.877)
  Change at Week 6: PAAP: number analyzed (Participants) | 40 | 26
  Change at Week 6: PAAP | -27.90 (20.061) | -12.35 (27.425)
  Change at Week 6: PGA: number analyzed (Participants) | 40 | 26
  Change at Week 6: PGA | -27.83 (18.936) | -11.65 (21.630)
  Change at Week 6: PGAA: number analyzed (Participants) | 40 | 26
  Change at Week 6: PGAA | -30.45 (17.868) | -19.50 (22.963)
  Change at Week 8: PAAP: number analyzed (Participants) | 39 | 24
  Change at Week 8: PAAP | -32.92 (25.051) | -18.58 (34.152)
  Change at Week 8: PGA: number analyzed (Participants) | 39 | 24
  Change at Week 8: PGA | -30.92 (21.279) | -15.88 (30.135)
  Change at Week 8: PGAA: number analyzed (Participants) | 39 | 24
  Change at Week 8: PGAA | -33.28 (18.725) | -23.75 (25.902)

18. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index [HAQ-DI] at Week 1, 2, 4, 6 and 8
Description: HAQ-DI assess degree of difficulty a participant experienced (during past week) in 8 domain of daily activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip and other activities. Each item scored on a 4-point scale ranging from 0 to 3(0=no difficulty; 3=extreme difficulty). Overall score: average of the sum of domain scores/number of domains answered. Total possible score range (0=least difficulty; 3=extreme difficulty); high scores=more difficulty in performing daily living activities.
Time Frame: Baseline, Week 1, 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-06651600 | Placebo
Number analyzed (Participants) | 42 | 28
units on a scale
  Baseline | 1.79 (0.577) | 1.69 (0.550)
  Change at Week 1: number analyzed (Participants) | 41 | 28
  Change at Week 1 | -0.13 (0.391) | -0.04 (0.316)
  Change at Week 2: number analyzed (Participants) | 42 | 27
  Change at Week 2 | -0.26 (0.430) | -0.15 (0.347)
  Change at Week 4: number analyzed (Participants) | 41 | 26
  Change at Week 4 | -0.39 (0.414) | -0.19 (0.534)
  Change at Week 6: number analyzed (Participants) | 40 | 26
  Change at Week 6 | -0.46 (0.527) | -0.23 (0.609)
  Change at Week 8: number analyzed (Participants) | 39 | 24
  Change at Week 8 | -0.53 (0.583) | -0.32 (0.671)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: Same event may appear as both an adverse event and serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | PF-06651600 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/28
Other Adverse Events (participants affected / at risk) | 20/42 | 5/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06651600 (N=42) | Placebo (N=28)
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 0
Oral herpes (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Cytomegalovirus test positive (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 3
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT02969044/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT02969044/SAP_001.pdf